CLINICAL TRIAL: NCT02666079
Title: A Multi-centre Clinical Study to Evaluate the LightPath® Imaging System in Wide Local Excision (WLE) for Breast Cancer
Brief Title: The LightPath® Breast Cancer Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lightpoint Medical Limited (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LPM-007
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Breast Cancer
Keywords: Wide local excision (WLE) for breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Wide local excision (WLE) for breast cancer with intra-operative use of the LightPath® Imaging System.
  Interventions: Device: LightPath® Imaging System.

INTERVENTIONS:
Device: LightPath® Imaging System. — Intra-operative use of the LightPath® Imaging System.

SUMMARY:
This study is a prospective, single arm, multi-centre study to evaluate the intra-operative use of the LightPath® Imaging System for the assessment of tumour margin status compared to hospital standard of care histopathology in wide local excision (WLE) for breast cancer

The intraoperative 18F-fluorodeoxyglucose (18F-FDG) LightPath® Images will be used to inform the surgeons about detectable residual cancer, in an attempt to achieve better guided cancer surgery and complete tumour excision with clear WLE resection margins.

Study sites will use the local criteria considered standard of care to guide decisions to act on positive margins.

In the LightPath® arm the resection margin status of the WLE specimen, cavity shavings (if any) and the metastatic status of axillary (sentinel) lymph nodes as measured with the LightPath® Imaging System will be compared with histopathology results.

DETAILED DESCRIPTION:
Female subjects with a diagnosis of invasive breast cancer scheduled to have wide local excision (WLE) +/- sentinel lymph node biopsy (SLNB) or axillary lymph node dissection (ALND) will be screened and receive 18F-FDG plus LightPath® Image. Subjects will have standard of care WLE. Extra cavity shaving due to positive 18F-FDG LightPath® Images is at the discretion of the surgeon.

Subjects will receive an intravenous injection of up to 5 MBq/kg, to a maximum 300 MegaBecquerel (MBq) of 18F-FDG prior to surgery.

Following resection, the WLE specimen will be examined using the LightPath® Imaging System. If the surgeons detect a positive signal they may perform cavity shavings of the resection cavity area corresponding to the positive signal area (up to a maximum thickness of 10mm).

Axillary SLNB will be performed according to local practice. At sites where 99mTc is used: In the 18F-FDG + LightPath® a higher dose of up to 150 MBq technetium-99m (99mTc) nanocolloid is necessary to avoid 18F-FDG masking the signal from 99mTc. Blue dye will be used according to local practice at sites where it is considered standard of care.

Sentinel lymph nodes (SLNs) will be examined using the LightPath® Imaging System. Where clinically indicated, ALND will be performed as per standard of care. At the time this protocol was finalised, LightPath® data involved lymph nodes sufficient to support recommendations were not available. For this reason, LightPath® Image results will not be used to direct ALND.

All LightPath® Images will be performed between 60 and 180 minutes post injection of 18F-FDG.

The WLE specimen, cavity shavings (where performed) and SLNs (where performed) will then undergo standard of care histopathological analysis. Lymph nodes will also be examined according to standard of care histopathological analysis. The results of the histopathological analysis will then be correlated with the LightPath® Images.

All staff in the operating room will wear badge dosimeters. Staff handling surgical specimens in theatre will also wear ring dosimeters. Histopathology analyses should be delayed to allow for radioactive decay of tissue samples to suitably low levels.

Subjects will be evaluated at screening and enrolment into the study. Data will be collected until the decision by the study site's MDT to recommend re-excision or mastectomy because of a positive margin on histopathological analysis (approx. 1-6 weeks post surgery)

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have signed an informed consent form prior to any study related activity
* Subjects who are able to give voluntary, written informed consent to participate in this study.
* Subjects who are able to understand this study and are willing to complete all the study assessments
* Female participants ≥18 years of age with a diagnosis of invasive breast cancer
* Subjects who have disease in one quadrant of the breast, not including the nipple
* Subjects scheduled for WLE for breast cancer +/- SLNB or ALND.
* Females of childbearing age must have a negative pregnancy test (by Beta human chorionic gonadotropin (HCG) qualitative analysis), or must have had a history of a surgical sterilisation, or must give history of no menses in the past twelve months

Exclusion Criteria:

* Subjects with pure DCIS or with pleomorphic LCIS
* Subjects who have had surgery in the ipsilateral breast in the past 12 months
* Subjects who have had radiotherapy in the ipsilateral breast
* Subjects who have had neoadjuvant systemic therapy
* Subjects who have had systemic chemotherapy in the past two years
* Subjects with a non-palpable lesion scheduled to have radio guided occult lesion localisation (ROLL)
* Subjects who have known hypersensitivity to 18F-FDG
* Subjects who are pregnant or lactating
* Subjects who have an existing medical condition that would compromise their participation in the study
* Subjects who have participated in a clinical study in the last 2 months
* Subjects with a current or active history of other known cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the LightPath® Imaging System | Initial surgery
  The diagnostic performance of tumour margin assessment with the LightPath® Imaging System compared to hospital histopathology.

SECONDARY OUTCOMES:
The recommendation by the study site's multidisciplinary team (MDT) to re-operate at the index location (breast) within 1 to 6 weeks post-initial surgery according to local practice. | 1-6 weeks post initial surgery
  MDT recommendation for the subject to undergo re-excision or mastectomy because of a positive margin on histopathological analysis.
Rate of re-operation at the index location | 1 to 6 weeks post initial surgery
  The number of subjects undergoing re-operation at the index location because of a positive margin on histopathological analysis, compared to published data on re-operation rates.
Volume of tissue excised | Initial surgery
  Weight (g) of all fresh pieces of tissue removed
Radiation dosimetry | Initial surgery
  Dosimetry readings will be summarised by staff member and procedure
Safety - adverse events (related to breast surgery) | Initial surgery
  Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether r not related to the device

OTHER OUTCOMES:
Agreement between LightPath® Image for lymph nodes status and histology | Initial surgery
  Proportion of lymph nodes that agree metastatic status
Biomarkers ER/PR/HER2 status | Screening
  ER/PR/HER2 will each be defined as positive or negative in accordance with local practice

CONTACTS AND LOCATIONS:
Overall Officials: Qamar B Akbar, MSc, Study Director — Clinical Project Manager
Locations (5):
- Poland (3):
  - Klinika Chirurgii Onkologicznej i Rekonstrukcyjnej Centrum Onkologii- Instytut oddział w Gliwicach, ul. Wybrzeże Armii Krajowej 15,, Gliwice
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Endokrynologii, ul. Mikołaja Kopernika 17,, Krakow
  - Centrum Onkologii - Instytut, im Marii Skłodowskiej-Curie, Klinika Nowotworów Piersi i Chirurgii Rekonstrukcyjnej ul. Roetgena 5, Warsaw
- United Kingdom (2):
  - Royal Liverpool Hospital, Liverpool
  - Cardiff Breast Centre, LLandough Hospital, Llandough

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jurrius PAGT, Grootendorst MR, Krotewicz M, Cariati M, Kothari A, Patani N, Karcz P, Nagadowska M, Vyas KN, Purushotham A, Turska-d'Amico M. Intraoperative [18F]FDG flexible autoradiography for tumour margin assessment in breast-conserving surgery: a first-in-human multicentre feasibility study. EJNMMI Res. 2021 Mar 18;11(1):28. doi: 10.1186/s13550-021-00759-w. PMID 33738563
- See also: Company website with description of the technology and Conformité Européenne (CE) marked medical device — http://www.lightpointmedical.com/
- See also: ISRCTN17778965 — http://www.isrctn.com/ISRCTN17778965